CLINICAL TRIAL: NCT05317910
Title: Evaluation of Effect of Music Therapy on Anxiety of Carers of Alzheimer's Disease Patients
Brief Title: Effect of Music Therapy on Anxiety of Caregivers of Alzheimer's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Musicothérapie Applications et Recherches Cliniques (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIDALZ
Record Dates: First submitted 2022-03-13; First posted 2022-04-08 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease
Keywords: Music intervention; Alzheimer; Anxiety
MeSH Terms: conditions — Alzheimer Disease; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music intervention (Experimental): Music intervention (duration 20 minutes) every day for 30 days
  Interventions: Other: MUSIC CARE

INTERVENTIONS:
Other: MUSIC CARE — Relaxation-type receptive musical intervention technique. The standardized 20-minute musical sequence is broken down into several phases that gradually lead the patient to relaxation using the new U-Mount technique [1, 2] (Figure 1). The effect works by reducing the musical rhythm, orchestral formation, frequencies and volume (the "U" descending phase). After a maximum relaxation phase (lower part of the "U"), a re-activating phase (ascending branch of the "U") is followed.

SUMMARY:
This clinical trial evaluates the impact of music interventions on caregivers of patients with memory disorders, Alzheimer's disease, dementia and related disorders. This study will follow caregivers of patients within the rehabilitation day care hospital "Memory and Frailty" (Hôpital de Jour de Réadaptation Mémoire et Fragilités), Sainte-Marie Paris Hospital.

DETAILED DESCRIPTION:
This clinical trial evaluates the impact of music on caregivers of patients with memory disorders, Alzheimer's disease, dementia and related disorders. This study will follow caregivers of patients within the rehabilitation day hospital "Memory and Frailty " (Hôpital de Jour de Réadaptation Mémoire et Fragilités), Sainte-Marie Paris Hospital.

All participants will benefit from a first session of a relaxation-type musical technique in the Day care Hospital (HDJ), they will then follow the sessions in their own homes. During the first visit, all participants will complete self-assessments, including a questionnaire on musical preferences and a self-assessment anxiety scale.

The expected inclusion period is 30 days. Carers will be equipped with tablets, headphones, eye masks and workbooks/questionnaires to use every day for one month in their homes. A relaxation-type receptive musical technique is used. The standardized 20-minute musical sequence is broken down into several phases that gradually lead the patient to a state of relaxation using the new U technique. The effect works by reducing the musical rhythm, orchestral formation, frequencies and volume (the "U" descending phase). After a maximum relaxation phase (lower part of the "U"), a re-activating phase (ascending branch of the "U") follows. All the musical sequences, built with the U-shape editing method, were specially produced by the music publishing company Music Care©. During the first session in HDJ, the subjects will lie on a relaxation table with a raised headrest (extended or semi-seated listening position) in an enclosed space, calm, secure and comfortable, with minimum lighting, so that the participant feels comfortable. The music will be played on headphones.

The main objective is to reduce anxiety among carers who accompany patients with memory disorders, Alzheimer's disease and related dementia.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety Self-Assessment Score (STAI) greater than 46 at Day 1
* Patient relationship (child, spouse, brother/sister)

Exclusion Criteria:

* Presence of a psychiatric disorder
* Intellectual disability
* Major hearing loss
* Professional musician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline STAI score at 28 days | Day 1 and Day 28
  Long-term anxiety will be measured using the State Trait Anxiety Inventory (STAI) scale. The STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Scores range from 20 to 80, with higher scores correlating with greater anxiety.

SECONDARY OUTCOMES:
Change on EVA score immediately after each session | Before and immediately after each session (up to 28 days (one session every day))
  Short-term anxiety will be evaluated by a Visual Analogue Scale (VAS) with a score from 0 to 10, which assesses caregiver anxiety, with higher scores correlating with greater anxiety.
Change from baseline STAI score at 15 days | Day 1 and Day 15
  Long-term anxiety will be measured using the State Trait Anxiety Inventory (STAI) scale. The STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Scores range from 20 to 80, with higher scores correlating with greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Marie Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided